CLINICAL TRIAL: NCT05915078
Title: Evaluation of Clinical and Health Economic Outcomes Following In-office Tympanostomy Using the Tula® System: a Prospective, Multi-center Registry
Brief Title: Evaluation of Outcomes Following In-office Tympanostomy Using the Tula® System: a Prospective, Multi-center Registry
Status: Recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Tula Registry
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media With Effusion; Acute Otitis Media; Otitis Media
Keywords: Otitis media; pediatric; tympanostomy; office procedure; local anesthesia
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media | interventions — Iontophoresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Tula Tympanostomy: Patients undergoing in-office tympanostomy using the Tula® System
  Interventions: Combination Product: Iontophoresis and tube placement

INTERVENTIONS:
Combination Product: Iontophoresis and tube placement — Iontophoretic delivery of TYMBION™ otic anesthetic using the Tula Iontophoresis System and tube insertion using the Tula Tube Delivery System

SUMMARY:
This prospective, single-arm, multicenter registry is being conducted to collect real world post-market data from patients aged from 6 months to 17 years of age who are undergoing an in-office ear tube placement procedure (tympanostomy) using the Tula® System. The Registry will include up to 20 centers in the US and up to 200 patients for the initial evaluation.

The FDA-approved Tula System includes the Tula Iontophoresis System (IPS) with TYMBION™ otic anesthetic for local anesthesia of the ear drum and the Tula Tube Delivery System (TDS) for ear tube placement. Clinical research established the safety, efficacy and tolerability of this system for in-office procedures in the pediatric population. Patients will be treated and evaluated according to standard medical care. Outcome data is collected up to 6 months following extrusion or removal of their tube(s).

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 6 months through 17 years of age (inclusive) at time of tympanostomy in-office using the Tula® System
* Patients who are candidates for in-office tube placement using the Tula System according to the System Instructions For Use

Exclusion Criteria:

* Patients who are wards are not included

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participating centers will invite eligible patients ages 6 months to 17 years of age indicated for tympanostomy to participate in the Registry
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Procedure Success | Day of procedure (day 0)
  Count (and percentage) of patients with successful placement of Tula Tympanostomy Tubes in all indicated ears in an office procedure

SECONDARY OUTCOMES:
Tolerability (physician reported) | Day of procedure (day 0)
  Count (and percentage) of patients that tolerated the procedure acceptably as determined by physician's observation.
Tolerability (parent reported) - anesthesia | Day of procedure (day 0)
  Count (and percentage) of patients whose parents strongly agree or agree with the statement 'My child tolerated the anesthesia process well'
Tolerability (parent reported) - procedure | Day of procedure (day 0)
  Count (and percentage) of patients whose parents strongly agree or agree with the statement 'The tube placement portion of the procedure was tolerable for my child'.
Recovery (physician reported) | Day of procedure (day 0)
  Count (and percentage) of patients who recovered once back with parent, or prior to leaving the clinic, following procedure completion as determined by physician's observation.
Recovery (parent reported) | Day of procedure (day 0)
  Count (and percentage) of patients who returned to normal activities immediately following the procedure.
Anesthesia effectiveness - patients | Day of procedure (day 0)
  Count (and percentage) of patients who completed iontophoresis with adequate anesthesia for tube placement in all treated ears as determined by the physician's evaluation of tympanic membrane anesthesia
Anesthesia effectiveness - ears | Day of procedure (day 0)
  Count (and percentage) of ears that completed iontophoresis with adequate anesthesia for TT placement as determined by the physician's tympanic membrane anesthesia evaluation.
Tula Tympanostomy Tube retention | 1 month post procedure
  Count (and percentage) of patients at the first post-operative visit in which a Tula Tympanostomy Tube was successfully placed, with presence of the Tula Tympanostomy Tube across the tympanic membrane
Parent satisfaction (informed) | 1 month post-procedure
  Count (and percentage) of patients whose parents strongly agree or agree with the survey question:
  'I felt well informed and prepared to help me/my child complete the procedure'
Parent satisfaction (siblings) | 1 month post-procedure
  Count (and percentage) of patients whose parents strongly agree or agree with the survey question:
  'If my child had a sibling who needed ear tubes, I would choose this procedure in the office instead of going under general anesthesia in the operating room'
Overall parent satisfaction | 1 month post-procedure
  Count (and percentage) of patients whose parents strongly agree or agree with the survey question:
  'Overall, I am very satisfied with the in-office ear tube procedure'
Parent satisfaction (recommendation) | 1 month post-procedure
  Count (and percentage) of patients whose parents strongly agree or agree with the survey question:
  'I would recommend this procedure to family/friends who have children who need ear tubes'

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Regional Otolaryngology Head and Neck Associates, Cherry Hill, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Columbia University Vagelos College of Physicians and Surgeons, New York, New York
  - Ogden Clinic - Professional Center North, Ogden, Utah
  - Peak Pediatric Ear, Nose and Throat, Provo, Utah